CLINICAL TRIAL: NCT03170661
Title: Effect of Deep Versus Moderate Neuromuscular Block During Sevoflurane Anesthesia on Intraoperative Surgical Conditions in Patients Undergoing Laparoscopic Renal Surgery
Brief Title: Effect of Deep Versus Moderate Neuromuscular Block During Sevoflurane Anesthesia on Intraoperative Surgical Conditions.
Acronym: BLISS4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Albert Dahan, Clinical professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: p17.049
Record Dates: First submitted 2017-04-25; First posted 2017-05-31 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Surgical Conditions
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate neuromuscular block (No Intervention): Subjects will receive moderate neuromuscular block, aimed at 1-2 twitches train of four
- Deep neuromuscular block (Experimental): Subjects will receive deep neuromuscular block, aimed at 1-2 twitches post tetanic count
  Interventions: Drug: Deep neuromuscular block

INTERVENTIONS:
Drug: Deep neuromuscular block — Deep neuromuscular block will be achieved with high dose rocuronium to achieve a depth of 1-2 twitches post tetanic count
  Other Names: high dose rocuronium
  Arms: Deep neuromuscular block

SUMMARY:
A deep neuromuscular block (NMB) is often associated with improved surgical conditions especially in laparoscopic surgery. We previously showed that deep NMB is superior to a moderate NMB under propofol anesthesia. However, this may not apply to sevoflurane anesthesia and sevoflurane by itself produces some degree of muscle relaxation. We therefore plan to investigate the effect of deep NMB on surgical conditions under sevoflurane anesthesia maintenance.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are routinely administered during general anaesthesia to facilitate endotracheal intubation and to optimize surgical conditions. Increasing data suggest superiority of a deep neuromuscular block (defined by a post-tetanic count of 1-2 twitches) in creating optimal working conditions for the surgical team. However, it is unknown whether other aspects of the anaesthetic technique, most notably the choice of anaesthetic (for example, total intravenous versus inhalational anaesthesia), influence the relationship between the depth of the neuromuscular block and surgical conditions, particularly in laparoscopic surgery. Volatile anaesthetics are known for their ability to potentiate neuromuscular blocking agents an effect that is less existent with propofol. We previously showed that surgical working conditions in laparoscopic surgery during propofol anaesthesia are highly reliant on the depth of the neuromuscular block. Whether such a relationship also exists for inhalational anaesthetics, is unknown. To investigate this, we conducted a prospective, randomized, double blind study in which patients scheduled for laparoscopic renal surgery were randomized to receive either a moderate or a deep neuromuscular block during sevoflurane anaesthesia. The primary outcome was the intraoperative surgical condition assessed by a surgeon using the validated Leiden-Surgical Rating Scale. We hypothesized that the use of an inhalational anaesthetic would obviate the need for a deep NMB due to its intrinsic muscle relaxant potentiating properties to produce optimal working conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with renal or prostatic disease who are will undergo an elective laparoscopic renal surgical procedure or laparoscopic prostatectomy;
* American Society of Anesthesiologists (ASA) class I-III
* > 18 years of age;
* Ability to give oral and written informed consent.

Exclusion Criteria:

* Known or suspected neuromuscular disorders impairing neuromuscular function;
* Allergies to muscle relaxants, anesthetics or narcotics;
* A (family) history of malignant hyperthermia;
* Women who are or may be pregnant or are currently breast feeding;
* Renal insufficiency, as defined by glomerular filtration rate < 30 ml/h creatinine.
* Previous retroperitoneal surgery at the site of the current surgery.
* Body mass index > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Started | 49 | 49
Completed | 49 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moderate Neuromuscular Block: Moderate neuromuscular block. In patients that were randomized to receive a moderate neuromuscular block, a bolus dose of rocuronium 0.5 mg kg-1 was administered, followed by intermittent injections of rocuronium 10-20 mg, aimed at keeping the train-of-four count at 1-2 twitches. At the end of the procedure, reversal of the neuromuscular block was by administration of sugammadex (2 mg kg-1). Patients were extubated when the train-of-four ratio reached 1.0, were breathing spontaneously and were awake.
- Deep Neuromuscular Block: In patients that were randomized to receive a deep neuromuscular block, a bolus dose of rocuronium 1.0 mg kg-1 was administered, followed by a continuous rocuronium infusion. The infusion rate was started at 0.3 mg kg-1 h-1 and titrated to keep the post-tetanic count at 1-2 twitches throughout the procedure. In case the surgeon scored Leiden-Surgical Rating Scale 1 or 2 (extremely poor or poor conditions), a bolus of rocuronium 10 mg could be administered. At the end of the procedure, reversal of the neuromuscular block was achieved with the administration of sugammadex 2-4 mg kg-1. Patients were extubated when the train-of-four ratio reached 1.0.
- Total: Total of all reporting groups
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Median (Full Range); unit: years] | 57 [20 to 77] | 51 [22 to 84] | 54 [20 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 21 | 20 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 49 | 49 | 98
Region of Enrollment [Number; unit: participants]
  Netherlands | 49 | 49 | 98
Procedure [Number; unit: Laparoscopic renal surgery] | 49 | 49 | 98
Height (m) [Mean (Standard Deviation); unit: m] | 1.75 (0.1) | 1.75 (0.1) | 1.75 (0.1)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 80 (13.5) | 81.4 (13.9) | 80.7 (13.7)
American Society of Anesthesiologists physical status classification system [Count of Participants; unit: Participants] — I A normal healthy patient II A patient with mild systemic disease III A patient with severe systemic disease IV A patient with severe systemic disease that is a constant threat to life V A moribund patient who is not expected to survive without the operation VI A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    1 | 22 | 28 | 50
    2 | 26 | 20 | 46
    3 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Leiden Surgical Rating Scale
Description: During the on average 3 hour procedure, the surgical condition will be scored by the surgeon using a 5-point surgical rating scale at 15 minute intervals(1: poor ; 5: optimal) Mean and standard deviation of the average of all leiden surgical rating scale will be reported.
Time Frame: during surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 49 | 49
score on a scale | 4.8 (0.4) | 4.8 (0.3)
Statistical Analysis 1: Comparison: Deep Neuromuscular Block; Test type: Superiority; p = 0.94, GEEGLM; Effects of GEEGLM covariates: surgeon, p = 0.24; surgery length, p= 0.73 and body mass index, p= 0.22)

2. Secondary Outcome: Postoperative Measurements and Outcomes; Pain Scores
Description: Postoperative measurements and outcomes of during PACU stay, all scores are reported as means and standard deviation of the average over the follow up period
  -mean pain scores (numeric rating scale; 0 no pain - 10 worst pain imaginable)
Time Frame: During post-anesthetic care unit stay (average stay 2 hours) at 15 minute intervals
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 49 | 49
units on a scale | 2.9 (1.9) | 3.2 (1.8)

3. Secondary Outcome: Intraoperative Hemodynamic Conditions
Description: Perioperative average blood pressure will be reported, mean blood pressure ranging from 65 tot 110 millimeters mercury is considered normal
Time Frame: Perioperative measurements at 15 minute interval (on average during 3 hours)
Measure: Median (Full Range); unit: millimeters mercury
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 49 | 49
millimeters mercury | 84 [67 to 103] | 85 [69 to 105]

4. Secondary Outcome: Postoperative Measurements and Outcomes; Sedation Levels
Description: Postoperative measurements and outcomes of during PACU stay, all scores are reported as means and standard deviation of the average over the follow up period
  -ramsay sedation levels (0 = normal alertness, eyes open, responds normal to command 1 = drowsy with open eyes, closed and opened on command 2 = drowsy with closed eyes, opened in response to light auditory stimulus 3 = eyes closed, opened in response to rubbing the shoulder or a loud auditory stimulus 4 = eyes closed and opened only briefly in response to touching the subject 5 = eyes closed, unarousable by touch, aroused by painful 6 = unarousable by pain)
Time Frame: During post-anesthetic care unit stay (average stay 2 hours) at 15 minute intervals
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 49 | 49
units on a scale | 0.9 (0.6) | 1.0 (0.6)

5. Secondary Outcome: Postoperative Measurements and Outcomes; Saturation
Description: Postoperative measurements and outcomes of during PACU stay, all scores are reported as means and standard deviation of the average over the follow up period
  -blood oxygen saturation in percent levels between 95-100 are considered normal
Time Frame: During post-anesthetic care unit stay (average stay 2 hours) at 15 minute intervals
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 49 | 49
percentage of blood oxygen saturation | 98 (1) | 98 (1)

6. Secondary Outcome: Intraoperative Nociception Level
Description: The median and full range of the average nociception level index will be reported.
  The nociception level index consist of Ta multiparameter nonlinear combination of heart rate, heart rate variability, amplitude of the finger photoplethysmogram, skin conductance level, fluctuations in skin conductance, and their time derivatives, derived from random forest regression. Random forest is an algorithmic modeling approach that enables combining multiple parameters of different origin and discovering their complex nonlinear interactions. Normal range is between 10-20; 0 indicates no nociceptive events (in example, pain stimuli), 100 indicates severe painful stimuli.
Time Frame: Perioperative measurements at 15 minute interval (on average during 3 hours)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 49 | 49
score on a scale | 11 [1 to 42] | 13 [4 to 27]

ADVERSE EVENTS:
Time Frame: Seven days post-procedure follow-up period
Description: The definition of adverse events is comparable to the definition by this website
Groups:
- Moderate NMB: Moderate neuromuscular block. In patients that were randomized to receive a moderate neuromuscular block, a bolus dose of rocuronium 0.5 mg kg-1 was administered, followed by intermittent injections of rocuronium 10-20 mg, aimed at keeping the train-of-four count at 1-2 twitches. At the end of the procedure, reversal of the neuromuscular block was by administration of sugammadex (2 mg kg-1). Patients were extubated when the train-of-four ratio reached 1.0, were breathing spontaneously and were awake.
- Deep NMB: In patients that were randomized to receive a deep neuromuscular block, a bolus dose of rocuronium 1.0 mg kg-1 was administered, followed by a continuous rocuronium infusion. The infusion rate was started at 0.3 mg kg-1 h-1 and titrated to keep the post-tetanic count at 1-2 twitches throughout the procedure. In case the surgeon scored Leiden-Surgical Rating Scale 1 or 2 (extremely poor or poor conditions), a bolus of rocuronium 10 mg could be administered. At the end of the procedure, reversal of the neuromuscular block was achieved with the administration of sugammadex 2-4 mg kg-1. Patients were extubated when the train-of-four ratio reached 1.0.
Arm/Group | Moderate NMB | Deep NMB
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 5/49 | 2/49
Other Adverse Events (participants affected / at risk) | 3/49 | 2/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate NMB (N=49) | Deep NMB (N=49)
prolonged hospital stay (Surgical and medical procedures) | 3 (3) | 2 (2)
hospital readmission (Surgical and medical procedures) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate NMB (N=49) | Deep NMB (N=49)
Postoperative CT-scan (Surgical and medical procedures) | 2 (2) | 1 (1)
Corneal Erosion (Surgical and medical procedures) | 0 (0) | 1 (1)
Reflex syncope (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03170661/Prot_SAP_000.pdf